CLINICAL TRIAL: NCT00565864
Title: Neurocognitive and Metabolic Effects of Mild Hypothyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Mary Samuels, Professor of Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00002265
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Hypothyroidism
Keywords: Hypothyroidism; Cognition; Metabolism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Low-normal TSH target) (Experimental): Treatment arm 1 targets a thyroid stimulating hormone (TSH) of 0.28 -2.49 milliunits/liter (mU/L) (the theoretical optimal range). The intervention is as follows: Levothyroxine (L-T4) doses will be adjusted in this arm to achieve this target TSH range. L-T4 is the intervention. L-T4 is given once per day, in the morning, while fasted. Dose ranges for the study are calculated based on each subject's TSH levels monitored during the study. Duration of the intervention is the duration of the study, after which subjects return to taking their usual L-T4 doses.
  Interventions: Drug: L-thyroxine (L-T4)
- 2 (High-normal TSH target) (Experimental): Treatment arm 2 targeting a TSH of 2.5 - 5.0 mU/L. The intervention is as follows:
  Levothyroxine (L-T4) doses will be adjusted in this arm to achieve this target TSH range. L-T4 is the intervention. L-T4 is given once per day, in the morning, while fasted. Dose ranges for the study are calculated based on each subject's TSH levels monitored during the study. Duration of the intervention is the duration of the study, after which subjects return to taking their usual L-T4 doses.
  Interventions: Drug: L-thyroxine (L-T4)
- 3 (Mildly elevated TSH target) (Experimental): Treatment arm 3 is targeting a TSH level o f 5.1-12.0 mU/L. The intervention is as follows:
  Levothyroxine (L-T4) doses will be adjusted in this arm to achieve this target TSH range. L-T4 is the intervention. L-T4 is given once per day, in the morning, while fasted. Dose ranges for the study are calculated based on each subject's TSH levels monitored during the study. Duration of the intervention is the duration of the study, after which subjects return to taking their usual L-T4 doses.
  Interventions: Drug: L-thyroxine (L-T4)

INTERVENTIONS:
Drug: L-thyroxine (L-T4) — L-thyroxine (L-T4) is the intervention for each arm/group. In each arm/group, the dose of L-T4 is adjusted to achieve TSH levels in the randomly assigned arm. L-thyroxine at doses appropriate to attain target TSH levels for the different arms for 24 weeks
  Other Names: Subjects will remain on their usual brand of L-T4.; Subjects on generic L-T4 will be switched to Levoxyl.

SUMMARY:
Patients with hypothyroidism are routinely treated with thyroid hormone (l-thyroxine) for replacement therapy. Physicians monitor the thyroid hormone dose by measuring a thyroid stimulating hormone (TSH) level in the blood, with the goal of a normal level. However, recent data suggest that the "normal" TSH range is too broad, and that patients may still have symptoms if their TSH levels are at the top or bottom part of the normal range.

To study this issue, it is useful to address issues such as general health status, psychological symptoms, mood, memory, and metabolic status, since thyroid hormone has major effects on the brain and metabolism, and since patients with treated hypothyroidism often have symptoms related to these areas.

In the present study, otherwise healthy subjects with treated hypothyroidism, ages 20-75 years, will be enrolled in a 7-11month study. At baseline, they will have tests of health status, psychological symptoms, mood, memory, body composition, and energy expenditure performed. Following these baseline measurements, subjects will receive either their usual doses of l-thyroxine, or a slightly higher or lower dose. The doses will be chosen to try to achieve either a low-normal TSH level, a high-normal TSH level, or a mildly elevated TSH level. Which target TSH the patient is assigned will be determined randomly, and neither the subject nor the study contacts will know which dose the patient is receiving. Subjects will be seen every 6 weeks during the study for brief visits to make sure they are not having any side effects, and to adjust the l-thyroxine doses if the TSH has not yet reached the target range. At the 24-week visit (end of study), the subjects will undergo the same tests that they had on the baseline visit.

Results from the study will be examined to see if minor changes in TSH or other thyroid hormone levels cause changes in any of the outcomes, and if the degree of TSH change correlates with the degree of outcome changes. These results may help physicians caring for patients with thyroid disease better determine the optimal dose of thyroid hormone for each patient.

DETAILED DESCRIPTION:
Thyroid hormone is essential for neurocognitive and metabolic function, and patients with overt thyroid dysfunction have well-described alterations in mood, cognition, energy expenditure, and body composition. However, it is not clear that patients with more mild degrees of thyroid dysfunction have clinically significant alterations in these parameters.

In addition, recent data suggest that variations in thyroid function within the laboratory reference range may also affect these parameters.

Patients with hypothyroidism are routinely treated with levothyroxine (L-T4) as replacement therapy. Physicians monitor the L-T4 dose by measuring serum thyroid stimulating hormone (TSH) levels, with the goal of a normal level. However, many patients with normal TSH levels continue to report symptoms, primarily in neurocognitive and metabolic areas. For this reason, patients with hypothyroidism often request higher L-T4 doses, but the clinical consequences of this are unknown.

In the present study, otherwise healthy subjects with treated hypothyroidism and normal TSH levels, ages 20-75 years, will be enrolled in a 7-11 month study. At baseline, the following tests will be performed to measure health status, psychological symptoms, mood, memory, body composition, and energy expenditure: the Short Form Health Survey-36 (SF-36), Profile of Mood States (POMS), Affective Lability Scale (ALS), Letter Cancellation Test (LCT), Trail Making Test, Iowa Gambling Task (IGT), N-Back Test, Subject-Ordered Pointing, Paragraph Recall, Pursuit Rotor, Motor Sequence Learning Test, resting energy expenditure (REE) and thermic effect of food (TEF) by indirect calorimetry, total energy expenditure (TEE) by doubly labelled water, physical activity energy expenditure (PAEE) by accelerometry, diet intake by 24-hour diet recalls, and body composition by dual energy x-ray absorptiometry (DEXA). Following these baseline measurements, subjects will receive either their usual doses of L-T4, or a slightly higher or lower dose. The doses will be chosen to try to achieve either a low-normal TSH level, a high-normal TSH level, or a mildly elevated TSH level. Which target TSH the patient is assigned will be determined randomly, and neither the subject nor the study contacts will know which dose the patient is receiving. Subjects will be seen every 6 weeks during the study for brief visits to make sure they are not having any side effects, and to adjust L-T4 doses if the TSH has not yet reached the target range. At the 24-week visit (end of study), the subjects will undergo the same tests that they had on the baseline visit.

Results from the study will be examined to see if minor changes in TSH or other thyroid hormone levels cause changes in any of the outcomes, and if the degree of TSH change correlates with the degree of outcome changes. These results may help physicians caring for patients with thyroid disease better determine the optimal dose of thyroid hormone for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20-75
* Primary hypothyroidism on stable dose of L-T4 for > 3 months
* Documented elevated TSH off L-T4
* Normal TSH level on usual dose of L-T4
* No acute or chronic medical or psychiatric illnesses that affect thyroid function, mood or cognition
* No medication use that affects thyroid function, mood or cognition (oral contraceptives or estrogen therapy allowed)
* Normal score on screening Mini-Mental State Exam (MMSE) (to test for dementia)
* Normal vision by screening examination
* Normal hearing by screening examination
* Non smoker

Exclusion Criteria:

* Failure to meet any of the above inclusion criteria
* Inability to speak and comprehend English
* A history of coronary artery disease
* Screening hgb <10
* Screening wbc > 10,000
* Clinically significant abnormalities on screening metabolic set
* Screening LDL cholesterol > 160
* Screening triglyceride > 300
* Significant abnormalities on screening ECG
* Pregnancy or intent to become pregnant in next 6 months
* Present or recent use of medications that affect thyroid hormone levels or interfere with thyroid hormone effects, including beta-blockers, lithium, glucocorticoids, or iodine containing agents
* MMSE score < 26

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2008-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Samuels, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Samuels MH, Kolobova I, Niederhausen M, Purnell JQ, Schuff KG. Effects of Altering Levothyroxine Dose on Energy Expenditure and Body Composition in Subjects Treated With LT4. J Clin Endocrinol Metab. 2018 Nov 1;103(11):4163-4175. doi: 10.1210/jc.2018-01203. PMID 30165520
- [Derived] Samuels MH, Kolobova I, Niederhausen M, Janowsky JS, Schuff KG. Effects of Altering Levothyroxine (L-T4) Doses on Quality of Life, Mood, and Cognition in L-T4 Treated Subjects. J Clin Endocrinol Metab. 2018 May 1;103(5):1997-2008. doi: 10.1210/jc.2017-02668. PMID 29509918
- [Derived] Samuels MH, Kolobova I, Antosik M, Niederhausen M, Purnell JQ, Schuff KG. Thyroid Function Variation in the Normal Range, Energy Expenditure, and Body Composition in L-T4-Treated Subjects. J Clin Endocrinol Metab. 2017 Jul 1;102(7):2533-2542. doi: 10.1210/jc.2017-00224. PMID 28460140
- [Derived] Samuels MH, Kolobova I, Smeraglio A, Niederhausen M, Janowsky JS, Schuff KG. Effect of Thyroid Function Variations Within the Laboratory Reference Range on Health Status, Mood, and Cognition in Levothyroxine-Treated Subjects. Thyroid. 2016 Sep;26(9):1173-84. doi: 10.1089/thy.2016.0141. Epub 2016 Jul 25. PMID 27338133
- [Derived] Samuels MH, Kolobova I, Smeraglio A, Peters D, Purnell JQ, Schuff KG. Effects of Levothyroxine Replacement or Suppressive Therapy on Energy Expenditure and Body Composition. Thyroid. 2016 Mar;26(3):347-55. doi: 10.1089/thy.2015.0345. Epub 2016 Feb 3. PMID 26700485
- [Derived] Samuels MH, Kolobova I, Smeraglio A, Peters D, Janowsky JS, Schuff KG. The effects of levothyroxine replacement or suppressive therapy on health status, mood, and cognition. J Clin Endocrinol Metab. 2014 Mar;99(3):843-51. doi: 10.1210/jc.2013-3686. Epub 2014 Jan 13. PMID 24423358

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Normal baseline thyroid stimulating hormone (TSH) Target TSH 0.28 - 2.50 milliunits/liter (mU/L)
- Arm 2: Normal baseline thyroid stimulating hormone (TSH) target TSH 2.51 - 5.60 milliunits/liter (mU/L)
- Arm 3: Normal baseline thyroid stimulating hormone (TSH) target TSH 5.61 - 12.0 milliunits/liter (mU/L)
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 58 | 59 | 56
Completed | 46 | 47 | 45
Not Completed | 12 | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Normal baseline TSH Target TSH 0.28 - 2.50 mU/L
- Arm 2: Normal baseline TSH target TSH 2.51 - 5.60 mU/L
- Arm 3: Normal baseline TSH target TSH 5.61 - 12.0 mU/L
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 46 | 47 | 45 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (11.5) | 50.9 (12.3) | 49.3 (10.7) | 49.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 43 | 125
  Male | 5 | 6 | 2 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 3 | 7
  Not Hispanic or Latino | 45 | 44 | 42 | 131
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 44 | 41 | 42 | 127
  More than one race | 0 | 3 | 1 | 4
  Unknown or Not Reported | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Executive Function
Description: Iowa Gambling Task Net-5. Four decks of cards are shown face down on a computer screen. The subject chooses cards from any deck, resulting in the gain or loss of money. The subject is unaware that 2 decks are advantageous (small gains, smaller losses), while 2 are disadvantageous (large gains, larger losses). The subject's choices are classified as advantageous (X) or disadvantageous (Y), with a net score of X-Y, over 5 trials of 100 cards each. The outcome reported here is the score on the fifth trial, which is generally the best trial due to practice effects. The minimum score is -20 and the maximum score is +20. Higher scores indicate a better outcome.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 46 | 47 | 45
units on a scale | 7.9 (1.6) | 7.5 (1.5) | 8.8 (1.6)

2. Primary Outcome: Resting Energy Expenditure
Description: Measurement of resting energy expenditure (REE) by indirect calorimetry, corrected for lean body mass. Indirect calorimetry is performed at 21.1° C after the participant has fasted for 12h and abstains from significant physical activity for 24h. The indirect calorimeter (VMax Encore 29N Indirect Calorimeter, SensorMedics Viasys Healthcare, Yorba Linda, CA) samples expired air and analyzes it for the volume of oxygen consumed (VO2) and the volume of carbon dioxide produced (VCO2) each minute for 30mins. REE is then calculated using the modified Weir equation. Minimum REE is 23 kcal/kg LBM/day and maximum REE is 39 kcal/kg LBM/day. Within that range, higher levels are considered better for the purposes of this study.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: kcal/kg LBM/day
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 46 | 47 | 45
kcal/kg LBM/day | 30.3 (0.4) | 30.0 (0.4) | 30.0 (0.5)

3. Other Pre Specified Outcome: Quality of Life by SF-36 Survey
Description: Short Form Survey (SF-36) mental component summary, which combines results from mental component subscales of the SF-36. The SF-36 health survey (SF-36) is a questionnaire about general health and well-being (127). It consists of 8 subscales (bodily pain, general health, mental health, physical functioning, vitality, role physical, social functioning, role emotional) and two summary scales (Mental Component and Physical Component Summaries). The mental component summary is a weighted average of the 8 subscales, with more weight to role emotional and mental health subscales. Minimum score for the SF-36 mental component summary is 14. Maximum score is 50. Higher scores on the SF-36 summary scales and subscales reflect better health status and well-being.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 46 | 47 | 45
units on a scale | 41.0 (0.9) | 39.8 (1.1) | 39.4 (1.0)

4. Other Pre Specified Outcome: Mood
Description: Profile of Mood States (POMS) fatigue subscale. The POMS consists of survey questions that cover 6 subscales: anxiety, confusion, depression-dejection, fatigue, tension, and vigor. Each subscale score is calculated from weighted averages of individual questions related to the subject's perception of fatigue. Minimum score for the fatigue subscale is 0. Maximum score is 30. Higher scores on the POMS fatigue subscale are worse.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 46 | 47 | 45
units on a scale | 7.4 (0.8) | 6.7 (0.9) | 6.9 (0.8)

5. Other Pre Specified Outcome: Working Memory
Description: 3-Back correct on target. The N-Back test consists of three conditions of increasing load on working memory, the 1-Back, 2-Back and 3-Back. In the 1-Back, letters are presented one at a time on a computer screen for 2 sec (1 sec interstimulus interval) during which the subject responds with a key press if a particular letter appears that had appeared on the previous screen. In the 2-Back, the subject must hold in mind letters and respond when s/he sees a letter that was previously presented two screens back. In the 3-Back, the subject responds when s'he sees a letter that was presented three screens back. N-back test measures the updating and storage functions of working memory. The test is scored as the number of targets correctly identified in each condition. The outcome of interest here is the number correct on target during the 3-Back, which is the most difficult of the three conditions. Minimum score is 0. Maximum score is 16. Higher scores are better.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 46 | 47 | 45
units on a scale | 11.7 (0.3) | 11.5 (0.4) | 11.5 (0.4)

6. Other Pre Specified Outcome: Declarative Memory
Description: Paragraph Recall - 30 min. Subjects were read a brief story and verbally recalled it immediately and after 30 minutes. The score was the total number of story elements recalled at 30 minutes. Minimum score is 0; Maximum score is 20. Higher scores are better.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 46 | 47 | 45
units on a scale | 11.9 (0.4) | 12.1 (0.5) | 12.8 (0.4)

7. Other Pre Specified Outcome: Motor Learning
Description: Pursuit Rotor Trial 4. This test is performed on a photoelectric pursuit Rotor (Model 30014, Lafayette Instrument Company, Lafayette, IN). Subjects hold a photosensitive wand to maintain contact with a 2 cm. light disk rotating on a variable speed turntable. An initial block of 4 trials is administered at 15, 30, 45, and 60 revolutions per minute. The speed at which the subject remains on-target is the rate at which remaining trials are performed. Three blocks of eight 20-second trials are then administered, with a 20-sec rest after each trial, and a 60-sec rest period after 4 trials. This sequence is repeated after a retention interval of 30 minutes. The measure of interest here is the time the wand maintains on target during the final trial. Minimum score is 0; maximum score is 80 seconds. Higher numbers are better.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 46 | 47 | 45
seconds | 41.8 (2.3) | 39.4 (1.9) | 45.0 (2.2)

8. Other Pre Specified Outcome: Total Energy Expenditure
Description: Total energy expenditure (TEE) measured by isotopic doubly labelled water (DLW) technique, corrected for lean body mass. A urine sample is collected and analyzed for background enrichment of deuterium and 18-O. The subject then drinks a dose of doubly labeled water at 1.7 gm per kg body weight, Samples are collected 2, 3 and 4 hours and seven days following the DLW dose to determine whole body equilibrium. Samples are measured as a ratio of deuterium to hydrogen in hydrogen gas and 18-O/ 16-O in CO2 using a Europa 20/20 Isotope Ratio Mass Spectrometer (Metabolic Solutions, Inc., Nashau, NH). CO2 production is then used to calculate TEE by Weir's equation. Minimum value is 36 kcal/kg LBM/day. Maximum value is 74 kcal/kg LBM/day. Within this range, higher values are considered to be better for the purposes of this study.
Time Frame: 24 weeks
Population: The number of participants analyzed is less than the total number of participants due to a nationwide shortage of doubly labelled water during the study. This meant that not all subjects entered into the study were able to receive the doubly labelled water.
Measure: Mean (Standard Error); unit: kcal/kg LBM/day
Arm/Group | Arm 2 | Arm 1 | Arm 3
Number analyzed (Participants) | 23 | 19 | 23
kcal/kg LBM/day | 53.0 (1.6) | 51.1 (1.5) | 50.6 (1.1)

9. Other Pre Specified Outcome: Thermic Effect of Food
Description: Thermic effect of food (TEF)is a measurement of energy expenditure over 5 hours following consumption of a standard test meal by indirect calorimetry. Each subject consumes a liquid mixed meal (Ensure, Ross Laboratories, 14% protein, 31.5% fat, and 54.5% carbohydrate) over 5 minutes and sampling for O2 and CO2 is then done by indirect calorimetry for the last 6 min of every 0.5 h for 5 h. For each metabolic measurement the respiratory exchange ratio (respiratory quotient or RQ = VCO2/VO2) is calculated and results converted to kilocalories by the Weir equation. Minimum value is 5 kcal/day. Maximum value is 730 kcal/day. Within this range, higher values are considered to be better for the purposes of this study.
Time Frame: 24 weeks
Population: The number of subjects who underwent measurement of thermic effect of food was less than the total number of subjects in the study due to scheduling constraints. TEF measurements take over 5 hours, and some subjects did not have sufficient time to participate in this part of the study, but were still able to conduct the other activities.
Measure: Mean (Standard Error); unit: kcal/day
Arm/Group | Arm 2 | Arm 1 | Arm 3
Number analyzed (Participants) | 26 | 23 | 31
kcal/day | 147 (28) | 136 (13) | 125 (12)

10. Other Pre Specified Outcome: Physical Activity Energy Expenditure
Description: Physical activity energy expenditure (PAEE) by accelerometry, corrected for lean body mass. The Actical activity monitoring device (Mini Mitter Co Inc, Bend, OR) utilizes a multidirectional accelerometer to monitor the occurrence and intensity of motion, or epoch (137). The Actical device measures 3 cm by 3 cm, weighs 17.0 grams, and is securely attached to a waistband and placed around the waist. The device is worn for 7 days. Data are downloaded from the accelerometer using an ActiReader and converted into total activity counts, average activity (counts per minute), time interval duration (minutes), activity ranges during sedentary, light, moderate, and vigorous activity, and accumulated time within each activity range (minutes). These data are then converted to PAEE by proprietary algorithms. Minimum value is 3 kcal/kg LBM/day. Maximum value is 40 kcal/kg LBM/day. Higher values are better.
Time Frame: 24 weeks
Population: A few subjects did not have data collected due to a technical problem with downloading their data from the Actical device.
Measure: Mean (Standard Error); unit: kcal/kg LBM/day
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 45 | 46 | 43
kcal/kg LBM/day | 11.6 (0.7) | 12.6 (0.6) | 11.4 (0.6)

11. Other Pre Specified Outcome: Daily Energy Intake
Description: Daily caloric intake is measured by 24-hour diet recalls, corrected for lean body mass (LBM). Three 24h food recall interviews are conducted by telephone within one week of the testing visit by research nutritionists trained in the Nutrition Data System for Research (NDSR), a software application for the collection of dietary recall information in a standardized fashion. Data from the phone interviews are manually entered into the NDSR program, which calculated caloric intake. The average of the three diet recalls is used as the outcome. Minimum value is 10 kcal/kg LBM/day. Maximum value is 72 kcal/kg LBM/day. Lower values are considered better for the purposes of this study.
Time Frame: 24 weeks
Population: One subject could not be reached by telephone to conduct the diet recalls.
Measure: Mean (Standard Error); unit: kcal/kg/day
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 46 | 47 | 44
kcal/kg/day | 26.8 (1.3) | 28.6 (1.6) | 27.4 (1.2)

12. Other Pre Specified Outcome: Body Mass Index
Description: Body mass Index (BMI) is calculated as the weight in kg divided by the (height in meters squared). Minimum value is 18 kg/m2. Maximum value is 50 kg/m2. For the purposes of this study, lower values are considered better.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 46 | 47 | 45
kg/m2 | 28.6 (0.8) | 27.3 (0.8) | 27.6 (1.0)

13. Other Pre Specified Outcome: Lean Body Mass
Description: Lean body mass (LBM) is measured by dual energy X-ray absorptiometry (DEXA). Measurements are made using a Hologic Discovery A Densitometer (Hologic, Inc., Bedford, MA). Proprietary algorithms calculate LBM from DEXA data. Minimum value is 28 kg. Maximum value is 71 kg. For the purposes of this study, higher values are considered better.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: kg
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 46 | 47 | 45
kg | 46.2 (1.1) | 45.0 (1.4) | 43.8 (1.3)

14. Other Pre Specified Outcome: % Fat Mass
Description: % fat mass is measured by dual energy X-ray absorptiometry (DEXA). Measurements are made using a Hologic QDR Discovery A Densitometer (Hologic, Inc., Bedford, MA). Proprietary algorithms calculate % fat mass from DEXA data. Minimum value is 20%. Maximum value is 56%. For the purposes of this study, lower values are considered better.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: percentage of total mass
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 46 | 47 | 45
percentage of total mass | 38.2 (1.0) | 36.4 (1.2) | 38.1 (1.1)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47 | 0/45
Other Adverse Events (participants affected / at risk) | 2/46 | 2/47 | 3/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=46) | Arm 2 (N=47) | Arm 3 (N=45)
medication error (Product Issues) | 2 (2) | 1 (1) | 2 (2) — medication delivered to wrong participant or wrong dose
symptoms (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) — two patients developed symptoms unrelated to study and withdrew

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No